CLINICAL TRIAL: NCT03585400
Title: Validation of the REPS Prediction Tool to Improve Quality of Perioperative Care
Brief Title: Validation of the REPS Prediction Tool
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2018P000264
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Residual Neuromuscular Blockade; Curarization, Postoperative Residual; Postoperative Respiratory Complication
Keywords: Neuromuscular Blockade Agents; Neuromuscular Blockade Reversal; Perioperative Care; Quality Improvement; Respiratory Complication
MeSH Terms: conditions — Delayed Emergence from Anesthesia | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study: Observational Study: Not Applicable for Observational Studies
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Observational Study: Not Applicable for Observational Studies

SUMMARY:
Neuromuscular blocking agents' (NMBA) use during surgery is associated with postoperative respiratory complications and increased risk of readmission to the hospital following ambulatory surgery. Residual neuromuscular block (rNMB) after surgery is difficult to identify. We have recently developed the REsidual neuromuscular block Prediction Score (REPS), that predicts the risk for postoperative rNMB. Our primary objective is now to assess the predictive ability of the REPS for respiratory complications within seven days following general anaesthesia. The secondary objective is to compare the predictive values of REPS and train-of-four (TOF)-ratio below 0.90 for respiratory complications.

DETAILED DESCRIPTION:
Residual neuromuscular blockade occurs in about 20-60% of patients and depends on compound and dose of NMBA reversal agent used. While on the one hand, NMBAs optimize surgical conditions and facilitate mechanical ventilation in patients with ventilator asynchrony, on the other hand, these agents have been associated with respiratory complications and increased risk of readmission after ambulatory surgery. A consensus in regard to guidelines and thresholds to define the optimal strategy to optimize surgical conditions is yet to be achieved. We have shown that utilization of non-depolarizing muscle relaxants and their reversal agents can be improved by dedicated quality improvement techniques. We have also recently developed the REPS, a tool that predicts postoperative rNMB.

This is a retrospective, observational, cohort study based on on-file hospital data from Beth Israel Deaconess Medical Center, Boston, Massachusetts.

The primary aim is to validate the dichotomized REPS (high-risk versus low-risk for rNMB which corresponds to a REPS >4 and <4, respectively) for the outcome of postoperative respiratory complications with BIDMC data. The investigators will utilize the pre-defined variables identified to predict residual neuromuscular blockade (REPS) at BIDMC.

The secondary aim is to compare the predictive values of the dichotomized REPS with dichotomized train-of-four (TOF)-ratio (low TOF-ratio versus high TOF ratio which corresponds to a TOF-ratio <0.9 and >=0.9, respectively) for respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Non-cardiac surgery
* General anesthesia with intermediate-acting NMBAs (atracurium, cisatracurium, vecuronium, or rocuronium)
* Extubated in the operating room
* PACU after surgery

Exclusion Criteria:

* American Society of Anesthesiology (ASA) Physical Status Classification of 5 or 6
* Did not receive neuromuscular blocking agents
* Missing last covariates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent non-cardiac surgery under general anesthesia with intermediate-acting NMBAs and are admitted to the Post-Anaesthesia Care Unit (PACU) after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 101510 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Respiratory Complications (PRC) | After extubation, up to 7 days after surgery
  PRC composite of invasive mechanical ventilation requirement within 7 postoperative days or immediate post-extubation desaturation (SpO2 <90%) within 10 minutes.

OTHER OUTCOMES:
Hospital Readmission | Up to 30 days after discharge
  Hospital readmission defined as any admission to BIDMC.
Hospital Length of Stay | During hospital stay, on average 4 days, and no longer than 1 year
  Hospital length of stay defined as the number of days elapsed from hospital admission to hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470
- [Background] Brueckmann B, Sasaki N, Grobara P, Li MK, Woo T, de Bie J, Maktabi M, Lee J, Kwo J, Pino R, Sabouri AS, McGovern F, Staehr-Rye AK, Eikermann M. Effects of sugammadex on incidence of postoperative residual neuromuscular blockade: a randomized, controlled study. Br J Anaesth. 2015 Nov;115(5):743-51. doi: 10.1093/bja/aev104. Epub 2015 May 2. PMID 25935840
- [Background] Kotake Y, Ochiai R, Suzuki T, Ogawa S, Takagi S, Ozaki M, Nakatsuka I, Takeda J. Reversal with sugammadex in the absence of monitoring did not preclude residual neuromuscular block. Anesth Analg. 2013 Aug;117(2):345-51. doi: 10.1213/ANE.0b013e3182999672. Epub 2013 Jun 11. PMID 23757472
- [Background] Intercontinental Marketing Services (IMS) Health, Multinational Integrated Data Analysis System (MIDAS), September 2010
- [Background] McLean DJ, Diaz-Gil D, Farhan HN, Ladha KS, Kurth T, Eikermann M. Dose-dependent Association between Intermediate-acting Neuromuscular-blocking Agents and Postoperative Respiratory Complications. Anesthesiology. 2015 Jun;122(6):1201-13. doi: 10.1097/ALN.0000000000000674. PMID 25919486
- [Background] Rudolph MI, Chitilian HV, Ng PY, Timm FP, Agarwala AV, Doney AB, Ramachandran SK, Houle TT, Eikermann M. Implementation of a new strategy to improve the peri-operative management of neuromuscular blockade and its effects on postoperative pulmonary complications. Anaesthesia. 2018 Sep;73(9):1067-1078. doi: 10.1111/anae.14326. Epub 2018 Jul 4. PMID 29974459
- [Background] Rudolph MI, Ng PY, Deng H, Scheffenbichler FT, Grabitz SD, Wanderer JP, Houle TT, Eikermann M. Comparison of a novel clinical score to estimate the risk of REsidual neuromuscular block Prediction Score and the last train-of-four count documented in the electronic anaesthesia record: A retrospective cohort study of electronic data on file. Eur J Anaesthesiol. 2018 Nov;35(11):883-892. doi: 10.1097/EJA.0000000000000861. PMID 30020144
- [Derived] Patrocinio MD, Shay D, Rudolph MI, Santer P, Grabitz SD, Xu X, Nabel S, Bose S, Eikermann M. REsidual Neuromuscular Block Prediction Score Versus Train-of-Four Ratio and Respiratory Outcomes: A Retrospective Cohort Study. Anesth Analg. 2021 Sep 1;133(3):610-619. doi: 10.1213/ANE.0000000000005363. PMID 33497061